CLINICAL TRIAL: NCT02873728
Title: Remote Ischemic Conditioning for Treatment of Chronic Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Sherutei Briut Clalit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SOR 265-16 CTIL
Record Dates: First submitted 2016-08-17; First posted 2016-08-19 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Leg Ulcer; Varicose Ulcer
Keywords: chronic ulcer; diabetic ulcer; venous ulcer; remote ischemic conditioning
MeSH Terms: conditions — Leg Ulcer; Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RIC (Experimental): In the study group, a blood pressure cuff will be inflated to 50 mmHg above systolic blood pressure while the performing investigator examines the radial pulse to ensure complete blood flow obstruction. Ischemia will be performed for 3 cycles of 5 min each and 10 min resting between cycles.
  Interventions: Procedure: Remote Ischemic Conditioning
- Control (Sham Comparator): In the control group, a blood pressure cuff will be inflated to 10 mmHg (Sham procedure) for 3 cycles of 5 min each and 10 min resting between cycles.
  Interventions: Other: Control

INTERVENTIONS:
Procedure: Remote Ischemic Conditioning — Creation of Brief 5 min Ischemia to upper limb using a Blood pressure cuff
  Arms: RIC
Other: Control — Puting blood pressure cuff on upper limb and inflating to 10mmhg for 5 min
  Arms: Control

SUMMARY:
The goals of this series of studies is to test the effect of RIC on chronic leg ulcers (Diabetic ulcers and venous ulcers) - and to improve the understanding of its biological mechanism. This is a prospective, double-blind, randomized, shame procedure-controlled study.

DETAILED DESCRIPTION:
After getting patients informed consent. Initial evaluation that includes: Venous and Arterial vascular evaluation, Medical past History including medications and surgeries Documentation of the chronic wounds by description and photography with scale.

Base line blood test for CBC, HbA1C, Electrolytes, Urea, Cr, Liver enzymes. IL 1 IL 6 VEGF NO CD34 Adenosine All patients will received the standard wound care in use by the staff of the chronic wound clinic. Care givers will be blinded as to the study allocation of each patient. Patients will be divided randomly into two equal groups. Pressure cuffs will be applied to both arms of all subjects. The cuffs will be inflated and deflated intermittently for three cycles of 5 minutes each. In the study group, the cuffs will be inflated to 50 mmHg above systolic blood pressure while the performing investigator examines the radial pulse to ensure complete blood flow obstruction. In the control group, inflation will be up to 10 mmHg only. The patients will be followed for 10 weeks.

During this period, they will be examined every 2 weeks (5 follow-up visits); and in each of these visits the above procedure will be repeated including blood collection before intervention and 24-48h after intervention.

In each visit a "blinded" physician will photograph with scale the wound and grade the granulation tissue covering the wound on a scale from 0 to 5.

The primary end point of the study is the number of healed wounds and wound area change among the two groups. Secondary outcomes will be the degree of granulation tissue and levels of IL 1 IL 6 VEGF NO CD34 Adenosine

ELIGIBILITY:
Inclusion Criteria:All patients presented to Chronic/Hard to heal wound clinic at Soroka University medical center and Sherutei Briut Clalit regional clinic.

Wound that did not heal under proper medical care for over two months.

Exclusion Criteria:Ulcers suspected or proven to be malignant tumors. Patients that are planned for vascular intervention within the next month Patients that are planned for amputation within the next month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Wound Healing | 8 weeks
  Wound closure

SECONDARY OUTCOMES:
Granulation | 8 weeks
  Change of granulation of wound according to granulation scale
Wound rea change | 8 weeks
  Change in % of wound area

OTHER OUTCOMES:
Biomarkers | 8 weeks
  Levels of IL 1 IL6 VEGF, NCD34, Adenosine

CONTACTS AND LOCATIONS:
Overall Officials: Eldad Silberstein, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

IPD SHARING:
Plan to Share IPD: Undecided